CLINICAL TRIAL: NCT02737072
Title: A Phase 1a/1b Study of CXCR4 Peptide Antagonist (LY2510924) Administered in Combination With the Anti-PD-L1 Antibody, Durvalumab (MEDI4736), in Advanced Refractory Solid Tumors
Brief Title: A Study of LY2510924 and Durvalumab in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16387; I2V-MC-CXAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor
Keywords: immuno-oncology
MeSH Terms: interventions — LY2510924; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 mg LY2510924 + 1500 mg Durvalumab (Experimental): 20 milligrams (mg) LY2510924 given subcutaneously (SQ) once daily in combination with 1500 mg durvalumab given intravenously (IV) on Day 1 of each cycle (28 days).
  Interventions: Drug: LY2510924; Drug: Durvalumab
- 30 mg LY2510924 + 1500 mg Durvalumab (Experimental): 30 mg LY2510924 given SQ once daily in combination with 1500 mg durvalumab given IV on Day 1 of each cycle (28 days).
  Interventions: Drug: LY2510924; Drug: Durvalumab
- 40 mg LY2510924 + 1500 mg Durvalumab (Experimental): 40 mg LY2510924 given SQ once daily in combination with 1500 mg durvalumab given IV on Day 1 of each cycle (28 days).
  Interventions: Drug: LY2510924; Drug: Durvalumab

INTERVENTIONS:
Drug: LY2510924 — Administered SQ
Drug: Durvalumab — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of chemokine (C-X-C Motif) receptor 4 (CXCR4) peptide antagonist LY2510924 and durvalumab for phase 1a and 1b in participants with advanced refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a: Have histologic or cytologic confirmation of advanced solid tumor
* Have at least 1 measurable lesion assessable using standard techniques by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
* Have adequate organ function
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have provided tissue from a newly obtained core or excisional biopsy of a tumor lesion or a recent biopsy defined by ≤3 years since last documented progression of disease
* Have an estimated life expectancy of ≥12 weeks, in the judgment of the investigator

Exclusion Criteria:

* Have a serious concomitant systemic disorder including human immunodeficiency virus (HIV), active hepatitis B virus (HBV), active HCV, active autoimmune disorder or disease requiring high dose of steroids

  * Have a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection or chronic diarrhea
  * Have evidence of interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity or active, noninfectious pneumonitis
  * Have an active infection requiring systemic therapy
* Have had prior therapy with an anti-programmed cell death 1 (PD-1), anti-PD-L1, anti-PD-L2, or anticytotoxic T lymphocyte-associated antigen-4 antibody
* Moderate or severe cardiovascular disease
* Have symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment
* Have received a live vaccine within 30 days before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

REFERENCES:
- See also: Click here for more information about this study: A Study of LY2510924 and Durvalumab in Participants With Solid Tumors — https://www.lillytrialguide.com/en-US/studies/solid-tumor/CXAD#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in 2 parts. Phase 1a of the study consisted of a dose-escalation assessment and Phase 1b of the study included 2 expansion arms. The study was terminated after the Phase 1a part was complete. A participant completed the study if they completed at least 1 cycle.
Period: Overall Study
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
Started | 3 | 3 | 3
Received at Least One Dose of Drug | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.33 (22.12) | 60.00 (7.55) | 48.33 (3.21) | 54.89 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 2 | 3 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as 1 of the following adverse events(AE) reported during the Phase 1a DLT observation period,if considered to be definitely,probably,or possibly related to either study regimen by the investigator;and fulfills any 1 of the following criterion using(NCI)CTCAE version(v)4.03:Grade4 immune-related AE,Grade4 non-laboratory AE,any CTCAE Grade ≥3 QT prolongation AE,≥Grade3 colitis or noninfectious pneumonitis irrespective of duration,Grade3 immune-related AE(excluding colitis,QT prolongation,or pneumonitis) that does not downgrade to Grade2 within 3 days after onset of event despite optimal medical management including systemic corticosteroids,or does not downgrade to ≤Grade 1 or baseline within 14 days,Grade2 pneumonitis that does not resolve to ≤Grade 1 within 3 days of the initiation of maximal supportive care,including corticosteroid therapy,Grade3 toxicity lasting an extended time despite optimal supportive care and there were also laboratory abnormalities criterion.
Time Frame: Cycle 1 (28 Days)
Population: All participants who received at least one of dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of LY2510924
Description: MTD was determined after the evaluation of Phase 1a portion of the trial. For Phase 1a, any DLT-equivalent toxicities observed in Cycle 2 and beyond were also be considered in dose escalation and determining MTD/recommended Phase 2 dose. See outcome measure number 1 for the DLT criterion.
Time Frame: Cycle 1 (28 Days)
Population: All phase 1a participants who received at least one dose of study drug.
Measure: Number; unit: milligram (mg)
Groups:
- All Phase 1a Participants: 20 mg LY2510924 + 1500 mg Durvalumab:
  20 milligrams (mg) LY2510924 given subcutaneously (SQ) once daily in combination with 1500 mg durvalumab given intravenously (IV) on Day 1 of each cycle (28 days).
  30 mg LY2510924 + 1500 mg Durvalumab:
  30 mg LY2510924 given SQ once daily in combination with 1500 mg durvalumab given IV on Day 1 of each cycle (28 days).
  40 mg LY2510924 + 1500 mg Durvalumab:
  40 mg LY2510924 given SQ once daily in combination with 1500 mg durvalumab given IV on Day 1 of each cycle (28 days).
Arm/Group | All Phase 1a Participants
Number analyzed (Participants) | 3
milligram (mg) | 40

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC [0-∞]) of LY2510924 When Co-Administered With Durvalumab
Description: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC [0-∞]) of LY2510924 when Co-Administered with Durvalumab
Time Frame: Cycle 1 Day 1: Predose, 0.5, 2, 4, 6, 8, 24-30 hours; Day 15: Predose, 0.5, 2, 4, 6, 8 hours
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour /milliliter (ng *h/mL)
Groups:
- 20 mg LY2510924 + 1500 mg Durvalumab: 20 milligrams (mg) LY2510924 given subcutaneously (SQ) in combination with 1500 mg durvalumab given intravenously (IV).
- 30 mg LY2510924 + 1500 mg Durvalumab: 30 mg LY2510924 given SQ in combination with 1500 mg durvalumab given IV.
- 40 mg LY2510924 + 1500 mg Durvalumab: 40 mg LY2510924 given SQ in combination with 1500 mg durvalumab given IV.
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
Number analyzed (Participants) | 3 | 3 | 3
nanogram*hour /milliliter (ng *h/mL)
  Day 1 | 3390 (33) | 3430 (17) | 7490 (57)
  Day 15: number analyzed (Participants) | 3 | 3 | 2
  Day 15 | 1960 (258) | 4320 (11) | NA (NA) — For n=2, only range 6210 - 170000 was calculated.

4. Secondary Outcome: Number of Participants With Anti-Durvalumab Antibodies When Administered in Combination With LY2510924
Description: Number of participants with treatment-emergent positive Anti-Durvalumab antibodies was summarized by treatment group.
Time Frame: Predose Cycle 1 Day 1 through 90 Day Post Treatment Follow Up (Up To 12 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Best Overall Response of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Best overall response of CR or PR was defined using RECIST v 1.1 criteria. CR was defined as the disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR was defined as ≥30% decrease in sum of diameter(SOD) of target lesions taking as reference the baseline sum diameter. PD was defined as ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference the smallest sum of the longest diameters recorded since treatment started and an absolute increase in sum diameter of ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR/total number of participants)*100.
Time Frame: Baseline through Measured Progressive Disease or Death (Up To 12 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
Number analyzed (Participants) | 3 | 3 | 3
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With CR, PR, or Stable Disease (SD) (Disease Control Rate [DCR])
Description: DCR: percentage of participants with CR, PR, or SD using RECIST v 1.1 criteria. CR: disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR: ≥30% decrease in sum of diameter (SOD) of target lesions taking as reference baseline sum diameter. PD: ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference smallest sum of longest diameters recorded since treatment started and an absolute increase in sum diameter ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. SD: neither sufficient shrinkage to qualify for PR nor increase to qualify for PD. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR+SD/total number of participants)*100.
Time Frame: Baseline through Measured Progressive Disease (Up To 12 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
Number analyzed (Participants) | 3 | 3 | 3
percentage of participants | 100 | 33.3 | 0

ADVERSE EVENTS:
Time Frame: Up To 14 months
Description: All participants who received at least one dose of study drug.
Arm/Group | 20 mg LY2510924 + 1500 mg Durvalumab | 30 mg LY2510924 + 1500 mg Durvalumab | 40 mg LY2510924 + 1500 mg Durvalumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg LY2510924 + 1500 mg Durvalumab (N=3) | 30 mg LY2510924 + 1500 mg Durvalumab (N=3) | 40 mg LY2510924 + 1500 mg Durvalumab (N=3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg LY2510924 + 1500 mg Durvalumab (N=3) | 30 mg LY2510924 + 1500 mg Durvalumab (N=3) | 40 mg LY2510924 + 1500 mg Durvalumab (N=3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (2) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (2)
Pyrexia (General disorders) | 1 (2) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated after the Phase 1a part was complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT02737072/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT02737072/SAP_001.pdf